CLINICAL TRIAL: NCT03015389
Title: Wide Area Transepithelial Sample Esophageal Biopsy Combined With Computer Assisted 3-Dimensional Tissue Analysis (WATS3D) For the Detection of High Grade Esophageal Dysplasia and Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: CDx Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: CDx 810
Record Dates: First submitted 2017-01-05; First posted 2017-01-10 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Barrett Esophagus; Esophageal Dysplasia; Esophageal Adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Barrett's associated esophageal dysplasia
  Interventions: Procedure: Diagnostic Test

INTERVENTIONS:
Procedure: Diagnostic Test — WATS3D brush biopsy

SUMMARY:
This is a multi-center, prospective, randomized study which will enroll patients undergoing endoscopic surveillance due to a history of histologically confirmed dysplasia. A member of the research team will approach a potential subject to discuss participation in the study, including background of the proposed study, inclusion and exclusion criteria, benefits and risks of the procedures and follow-up. If this is of interest to the subject, the informed consent form is discussed and presented. The subject must sign the consent form prior to enrollment. This form will have prior approval of the study site's Institutional Review Board (IRB). Failure to obtain informed consent renders the subject ineligible for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age: ≥ 18 years
2. Patients should have a history of Barrett's associated esophageal dysplasia (either low or high-grade) confirmed on histology
3. Willingness to undergo both WATS3D and random forceps biopsies while undergoing conventional EGD with sedation
4. Ability to provide written, informed consent (approved by IRB) and understand the responsibilities of trial participation
5. Only patients who no visible mucosal abnormalities at the time that they undergo both random forceps biopsies and WATS3D testing of the esophagus will be included in this study

Exclusion Criteria:

1. Coagulopathy with INR > 2.0, thrombocytopenia with platelet counts < 50,000
2. The subject is pregnant or planning a pregnancy during the study period
3. History of esophageal or gastric surgery other than Endoscopic Mucosal Resection (EMR)
4. Patients who have undergone endoscopic ablative therapies
5. Subject has a known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions, or follow-up guidelines
6. Study patients with inadequate WATS3D specimens will not undergo a repeat brush biopsy test and will be excluded from the study
7. BE length < 1 cm or > 10 cm
8. Patients within six weeks of receiving targeted forceps biopsies and/or EMR
9. Patients with visible mucosal abnormality at the time of the WATS3D and random biopsy testing
10. Patients with visible lesions that are either submucosal or covered with a clinically intact epithelium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Barrett's associated esophageal dysplasia
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Detection rate of Barrett's associated high grade esophageal dysplasia and esophageal adenocarcinoma (HGD/EAC) using WATS3D and random 4 quadrant forceps biopsies taken at 2 cm intervals. | up to 2 years

SECONDARY OUTCOMES:
Number of participants with Barrett's related dysplasia and adenocarcinoma diagnosed with random forceps biopsies and WATS3D biopsies used in alternating fashion. | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Raf Bisschops, MD, Principal Investigator — University Hospitals Leuven, Dept. of Gastroenterology; Cesare Hassan, MD, Principal Investigator — Nuovo Regina Margherita Hospital
Locations (1):
- UZ Leuven - Campus Gasthuisberg, Leuven, Belgium